CLINICAL TRIAL: NCT04942951
Title: The Impact of Urinary Incontinence on Anxiety Status in Pregnancy Period: A Prospective Case-control Study
Brief Title: Urinary Incontinence and Anxiety in Pregnancy
Status: Completed | Type: Observational
Sponsor: Esin Merve Erol Koç (Other)
Responsible Party: Sponsor-Investigator, Esin Merve Erol Koç, Medical Doctor, Ankara City Hospital Bilkent
Organization: Ankara City Hospital Bilkent (Other)
Other Study IDs: 0067/2019
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Anxiety in Pregnancy (Disorder); Urinary Incontinence; Quality of Life
MeSH Terms: conditions — Urinary Incontinence | interventions — Gynecological Examination; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women with the diagnosis of urinary incontinence (Study group): The pregnant women who were diagnosed with the urinary incontinence (n=80) with category 0 or category 1 Pelvic Organ Prolapse Quantification (POP-Q) score in physical examination.
  Interventions: Diagnostic Test: Gynecological examination; Other: Pelvic Organ Prolapse Quantification (POP-Q); Other: Incontinence Consultation Questionnaire-Short Form (ICIQ-SF) questionnaire; Other: Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2) questionnaire
- Healthy pregnant women (Control group): Control group consisted of healthy women with uncomplicated pregnancies (n=80). They had no complaint of urinary incontinence and their gynecological examination did not reveal any finding of pelvic organ prolapse.
  Interventions: Diagnostic Test: Gynecological examination; Other: Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2) questionnaire

INTERVENTIONS:
Diagnostic Test: Gynecological examination — Gynecological examination was performed to the whole pregnant cohort included in the study to diagnose either the pelvic organ prolapse according to the POP-Q system or to be sure that they have no findings of pelvic organ prolapse.
Other: Pelvic Organ Prolapse Quantification (POP-Q) — Gynecological examination was performed to the whole pregnant cohort included in the study to diagnose either the pelvic organ prolapse according to the POP-Q system or to be sure that they have no findings of pelvic organ prolapse.
  Groups: Pregnant women with the diagnosis of urinary incontinence (Study group)
Other: Incontinence Consultation Questionnaire-Short Form (ICIQ-SF) questionnaire — ICIQ-SF questionnaire was applied to the Study group to determine the severity of urinary incontinence.
  Groups: Pregnant women with the diagnosis of urinary incontinence (Study group)
Other: Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2) questionnaire — PRAQ-R2 questionnaire was applied to the whole pregnant cohort included in the study to determine their anxiety status.

SUMMARY:
This prospective case-control study aimed to evaluate the impact of presence, and severity of urinary incontinence (UI) on pregnancy related anxiety. The study included 160 pregnant women with uncomplicated pregnancies at the second trimester. The pregnant women with UI (n=80) were compared to the control group including continent pregnant women (n=80) in terms of Pregnancy-Related Anxiety Scores (PRAQ-R2) and Incontinence Consultation Questionnaire-Short Form (ICIQ-SF) in pregnant women. Pelvic Organ Prolapse Questionnaire (POP-Q) was considered for the diagnosis of pelvic organ prolapsus. The UI was also divided into subgroups as stress (SUI), urge (UUI), and mixed (MUI) types and they were also compared to the control group.

DETAILED DESCRIPTION:
In this study, we aimed to evaluate the impact of the presence and the severity of UI on pregnancy related anxiety status in a well-defined pregnant cohort. The correlations were also analyzed in terms of the UI subtypes as stress urinary incontinence (SUI), urge urinary incontinence (UUI) and mixed urinary incontinence (MUI). A total of 160 pregnant women applied to outpatient clinics of Obstetrics and Urology Departments were included in the current study. Patients were compared in two groups in terms of Study group including pregnant women who were diagnosed with the UI (n=80) and Control group including healthy pregnant women (n=80). The study was approved by the institutional review board of Ankara Training and Research Hospital (# 0067/2019). All the participants were informed, and written consent was obtained before the participated the study.

Physical examination was performed to diagnose the pelvic organ prolapse and the findings were classified through the five categories based on Pelvic Organ Prolapse Quantification (POP-Q). According to POP-Q, only the pregnant women diagnosed with category 0 or category 1 were included in the study. All the pregnant women included in the current study were married and multiparous women, at the second trimester of the pregnancy, with uncomplicated pregnancies and regular pregnancy follow-up. Pregnancies complicated by chronic maternal diseases (rheumatological diseases, renal failure, vascular malformations, hypertension, cardiac disease, diabetes mellitus, obesity, hypo-hyperthyroidy, congenital hematological disorders), acute inflammatory conditions (acute pancreatitis, acute appendicitis), pregnancy complications (gestational diabetes, preeclampsia, preterm labor, preterm premature rupture of membranes), history of alcohol consumption, having multiple pregnancies, psychiatric diseases, cognitive disorders, neurogenic bladder, fecal incontinence, chronic constipation, chronic cough, urinary infection, history of pelvic surgery including incontinence surgeries and/or taking medication for UI were excluded from the current study. Pregnancy-Related Anxiety Questionnaire-Revised (PRAQ-R2) scale was used to evaluate the anxiety status of the participants. The International Consultation of Incontinence Questionnaire - Short Form (ICIQ-SF) which has been defined by Hajebrahimi et al. as a reliable scale, and validated in Turkish by Demircan et al. was used for the evaluation of UI. This scale includes questions about the frequency of UI, the conditions at which UI occurs and how much it affects the social life of the person. UI subtypes were diagnosed according to the definitions of the International Continence Society.

ELIGIBILITY:
Inclusion Criteria:

The pregnant women who were diagnosed with the urinary incontinence (n=80) with category 0 or category 1 Pelvic Organ Prolapse Quantification (POP-Q) score in physical examination.

Healthy women with uncomplicated pregnancies (n=80) with no complaint or finding of urinary incontinence.

Married and multiparous women, at the second trimester of the pregnancy, with uncomplicated pregnancies and regular pregnancy follow-up.

Exclusion Criteria:

Pregnancies complicated by chronic maternal diseases, acute inflammatory conditions, pregnancy complications, history of alcohol consumption, having multiple pregnancies, psychiatric diseases, cognitive disorders, neurogenic bladder, fecal incontinence, chronic constipation, chronic cough, urinary infection, history of pelvic surgery including incontinence surgeries and/or taking medication for urinary incontinence were excluded.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Study group: The pregnant women who were diagnosed with the urinary incontinence (n=80) with category 0 or category 1 Pelvic Organ Prolapse Quantification (POP-Q) score in physical examination.
  Control group: Consisted of healthy women with uncomplicated pregnancies (n=80). They had no complaint of urinary incontinence and their gynecological examination did not reveal any finding of pelvic organ prolapse.
  The pregnant women included both in the Study and Control group were married and multiparous women, at the second trimester of the pregnancy, with uncomplicated pregnancies and regular pregnancy follow-up.
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-06-05 (Actual)

PRIMARY OUTCOMES:
Pelvic Organ Prolapse Quantification (POP-Q) | 10 minutes
  graded between 0-4.

SECONDARY OUTCOMES:
Pregnancy-Related Anxiety Questionnaire-Revised 2 (PRAQ-R2) | 20 minutes
  scored between 10-50 points.

OTHER OUTCOMES:
Incontinence Consultation Questionnaire-Short Form (ICIQ-SF) | 20 minutes
  scored between 1-21 points.

CONTACTS AND LOCATIONS:
Overall Officials: Esin Merve Erol Koç, MD, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Esin Merve Erol Koç, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data will be available if needed by the review board.

REFERENCES:
- [Result] Felde G, Ebbesen MH, Hunskaar S. Anxiety and depression associated with urinary incontinence. A 10-year follow-up study from the Norwegian HUNT study (EPINCONT). Neurourol Urodyn. 2017 Feb;36(2):322-328. doi: 10.1002/nau.22921. Epub 2015 Nov 20. PMID 26584597
- [Result] Huizink AC, Delforterie MJ, Scheinin NM, Tolvanen M, Karlsson L, Karlsson H. Adaption of pregnancy anxiety questionnaire-revised for all pregnant women regardless of parity: PRAQ-R2. Arch Womens Ment Health. 2016 Feb;19(1):125-32. doi: 10.1007/s00737-015-0531-2. Epub 2015 May 14. PMID 25971851
- [Result] Hajebrahimi S, Corcos J, Lemieux MC. International consultation on incontinence questionnaire short form: comparison of physician versus patient completion and immediate and delayed self-administration. Urology. 2004 Jun;63(6):1076-8. doi: 10.1016/j.urology.2004.01.005. PMID 15183953
- [Result] Felde G, Bjelland I, Hunskaar S. Anxiety and depression associated with incontinence in middle-aged women: a large Norwegian cross-sectional study. Int Urogynecol J. 2012 Mar;23(3):299-306. doi: 10.1007/s00192-011-1564-3. Epub 2011 Nov 9. PMID 22068320